CLINICAL TRIAL: NCT04320108
Title: The Effects of Extracorporeal Shockwave Therapy (ESWT) for Shoulder Pain in Patients With Brain Damage
Brief Title: ESWT for Shoulder Pain in Patients With Brain Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principal professor of Rehabilitation Medicine, Bundang CHA Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESWTbraindamage
Record Dates: First submitted 2020-03-21; First posted 2020-03-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Brain Damage, Hypoxic; Stroke; Brain Tumor; ICH
Keywords: Extracorporeal shockwave therapy; Brain damage; Pain
MeSH Terms: conditions — Hypoxia, Brain; Stroke; Brain Neoplasms; Brain Injuries; Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): 3,000 pulses per time, low energy under 0.3 mJ/mm^2, tolerable range
  Interventions: Device: Extracorporeal shockwave therapy
- Control group (Sham Comparator): Sham therapy
  Interventions: Device: Extracorporeal shockwave therapy

INTERVENTIONS:
Device: Extracorporeal shockwave therapy — Extracorporeal shockwave therapy 6 times during 2 weeks

SUMMARY:
This study aimed to investigate the efficacy and safety of extracorporeal shockwave therapy (ESWT) for upper extremity pain related to spasticity in patients with spinal cord injury.

DETAILED DESCRIPTION:
6 times of ESWT (3,000 pulses per time, low energy under 0.3 mJ/mm^2, tolerable range) on subscapularis and lesser and greater tuberlces of humerus to reduce pain in patients with brain damage

ELIGIBILITY:
Inclusion Criteria:

* Brain damaged patient confirmed in the brain image
* 1 month after brain damage
* Pain in hemiplegic shoulder areas more than 4 points on the numerical scale (NRS)
* Cognitive functions that can clearly point out NRS with more than 15 points in the mini mental state examination (MMSE)
* Age: 20 and older
* Person who has agreed in writing to decide his or her participation and comply with the precautions

Exclusion Criteria:

* Pain due to trauma
* Injection treatments two weeks before participating in the study
* Severe coagulopathy (excluding antiplatelet use)
* Impaired cognition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Up to 4 weeks (baseline, after each treatment during 2 weeks, 2 weeks + 1 day, 4 weeks)
  Pain intensity (0-10, ordinal scale)

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Up to 4 weeks (baseline, 2 weeks + 1 day, 4 weeks)
  Scoring scale consist of 5 pain scale and 8 disability scale, in %, 0 (best) to 100 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, CHA Bundang Medical Center, CHA University School of Medicine
Locations (1):
- Department of Rehabilitation Medicine, CHA Bundang Medical Center, Seongnam, South Korea, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol